CLINICAL TRIAL: NCT06956638
Title: Predictors of Appendiceal Perforation and the Role of Total Bilirubin at Presentation: A Single Center Prospective Cross-sectional Study in Nepal
Brief Title: Bilirubin Levels to Diagnose Appendicitis and Predict Appendiceal Perforation
Status: Completed | Type: Observational
Sponsor: Nepalese Army Institute of Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB604
Record Dates: First submitted 2025-04-24; First posted 2025-05-04 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Acute Appendicitis; Appendicitis Perforated
Keywords: Single-center; prospective; cross-sectional
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients of age group above 5 years with acute appendicitis undergoing appendectomy: Patients of age group above 5 years with acute appendicitis undergoing appendectomy, without acute or chronic liver diseases, acquired or congenital bilirary diseases, history of use of hepatotoxic drugs or diagnosis of appendicular lump
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — Non-interventional study

SUMMARY:
The goal of this study is to learn if serum bilirubin levels can aid in the diagnosis of acute appendicitis and predict appendiceal perforation

DETAILED DESCRIPTION:
The study aims to assess hyperbilirubinemia: serum direct, indirect and total bilirubin to enhance the diagnostic accuracy of acute appendicitis. Also it aims to analyze different patient variables such as age, gender, duration of symptoms, leukocyte and neutrophil count, Alvarado score, presence of fever, nausea & vomiting, peritonitis alongside serum total bilirubin level in patients with appendicitis and assess which variables can be taken as independent factors to predict appendiceal perforation.

ELIGIBILITY:
Inclusion Criteria:

* Patients of age group above 5 years with acute appendicitis undergoing appendectomy with written informed consent.

Exclusion Criteria:

* Patients with appendicular lump.
* Patients with acute and chronic liver diseases like acute hepatitis, hemolytic disease, Gilbert's syndrome, Dubin-Johnson syndrome, alcoholic liver disease.
* Acquired or Congenital Biliary Disease.
* History of Hepatotoxic drugs.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients presenting with acute appendicitis at Shree Birendra Hospital, Chhauni, Kathmandu
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2022-07-16 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2025-03-12 (Actual)

PRIMARY OUTCOMES:
Perforated appendix | Presentation to hospital till perioperative period
  Perforated appendicitis was confirmed intraoperatively by the surgeon and at histological analysis of the specimen by the rupture of appendiceal wall to the serosa. Those with gangrenous walls were also taken as perforated.

CONTACTS AND LOCATIONS:
Overall Officials: Bhairav Kumar Hamal, MS, Fellow - Urosurgery, Study Chair — Nepalese Army Institute of Health Sciences
Locations (1):
- Shree Birendra Hospital, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Result] Sirikurnpiboon S, Amornpornchareon S. Factors Associated with Perforated Appendicitis in Elderly Patients in a Tertiary Care Hospital. Surg Res Pract. 2015;2015:847681. doi: 10.1155/2015/847681. Epub 2015 Aug 24. PMID 26380377
- [Result] Potey K, Kandi A, Jadhav S, Gowda V. Study of outcomes of perforated appendicitis in adults: a prospective cohort study. Ann Med Surg (Lond). 2023 Mar 16;85(4):694-700. doi: 10.1097/MS9.0000000000000277. eCollection 2023 Apr. PMID 37113955
- [Result] Chaudhary P, Kumar A, Saxena N, Biswal UC. Hyperbilirubinemia as a predictor of gangrenous/perforated appendicitis: a prospective study. Ann Gastroenterol. 2013;26(4):325-331. PMID 24714371
- [Result] Sand M, Bechara FG, Holland-Letz T, Sand D, Mehnert G, Mann B. Diagnostic value of hyperbilirubinemia as a predictive factor for appendiceal perforation in acute appendicitis. Am J Surg. 2009 Aug;198(2):193-8. doi: 10.1016/j.amjsurg.2008.08.026. Epub 2009 Mar 23. PMID 19306980
- See also: Related Info — https://bmcgastroenterol.biomedcentral.com/articles/10.1186/s12876-021-01614-x